CLINICAL TRIAL: NCT02154204
Title: A Validation Study of Near Infrared Fluorescence Imaging of Lymphatic Vessels in Humans.
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: NIRF2014
Record Dates: First submitted 2014-05-23; First posted 2014-06-03 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2014-05

CONDITIONS: Focus of Study is: Near Infrared Fluorescence Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The aim of this study is to examine the use of Near Infrared Fluorescence imaging on lymphatic vessels in humans.

Different parameters that reflect lymphatic function will be tested for intra and inter individual reproducibility.

We use 10 healthy test subjects and examine their lymphatic system. All subjects are healthy men between the ages of 20 and 30.

When the fluorescent dye "indocyanine green", has been injected into the skin on the patients feet, it will be transported through the lymph vessels, resulting in clear visualization of the vessels, using a laser and a EM-CCD camera.

On both legs we examine the frequency of vessel contraction and the velocity of lymph moving in vessels. We furthermore use several methods to quantify the vessel function such as the refill time of a vessel, (manually emptied vessel and refill time of 10 cm of a vessel), and pumping pressure (at what pressure lymph can pass a blood pressure cuff).

We investigate the activity of vessels over time, and after several interventions such as exercise, and water baths of the foot at different temperatures.

The patients are examined for approximately 4 hours and wil be examined again 14 days later.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* lymphedema, edema or vascular disease.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participants are young healthy males.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Frequency of contraction in lymph vessels. | At baseline and after 14 days
Pumping pressure | At baseline and after 14 days
refill time | At baseline and after 14 days
velocity | At baseline and after 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke E Hjortdal, MD, PhD, DMSc, Study Director — Department of cardiothoracic and vascular surgery, Aarhus university hospita; Jacob H Grønlund, bac. med., Principal Investigator — Department of cardiothoracic and vascular surgery, Aarhus university hospita
Locations (1):
- Department of cardiothoracic and vascular surgery, Aarhus university hospital., Aarhus N, Denmark